CLINICAL TRIAL: NCT05409287
Title: Influence of the Implant Loading Protocol on Implant Survival in Early Placed Single-tooth Implants in Mandibular Posterior Sites Using Computer-assisted Implant Surgery: A Randomized Clinical Trial (RCT)
Brief Title: Immediate Loading in Single Tooth Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITI 1400_2019
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Partial Edentulism Class 3
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Implant Loading (Experimental): A provisional single implant crown will be mounted on an implant, placed 16 weeks post tooth extraction, immediately after implant placement. Occlusion will be adjusted, so that there is no occlusal contact with the 8 µm Shim Stock foil (Hanel Shim Stock Foil; Coltène/Whaledent AG, Altsätten, Switzerland), but contact with 40µm occlusion foil (Hanel Articulating Paper, Coltène/Whaledent AG, Altsätten, Switzerland) during static occlusion. All dynamic contacts will be eliminated by intraoral grinding with a diamond bur, and the occlusal surface will be polished afterward. The screw access channel will be sealed by a Teflon strip and a provisional light-polymerizing resin (Telio CS, Ivoclar Vivadent AG, Schaan, Liechtenstein). In case of a mini-flap on the buccal aspect, the flaps will then be sutured around the implant healing cap or the implant provisional with single interrupted sutures. Finally, a periapical radiograph will be taken, using the customized x-ray tray.
  Interventions: Procedure: Immediate Implant Loading
- Early Implant Loading (Active Comparator): A provisional single implant crown will be mounted on an implant, placed 16 weeks post tooth extraction, 4 weeks after implant placement. Occlusion will be adjusted, so that there is no occlusal contact with the 8 µm Shim Stock foil (Hanel Shim Stock Foil; Coltène/Whaledent AG, Altsätten, Switzerland), but contact with 40µm occlusion foil (Hanel Articulating Paper, Coltène/Whaledent AG, Altsätten, Switzerland) during static occlusion. All dynamic contacts will be eliminated by intraoral grinding with a diamond bur, and the occlusal surface will be polished afterward. The screw access channel will be sealed by a Teflon strip and a provisional light-polymerizing resin (Telio CS, Ivoclar Vivadent AG, Schaan, Liechtenstein). In case of a mini-flap on the buccal aspect, the flaps will then be sutured around the implant healing cap or the implant provisional with single interrupted sutures. Finally, a periapical radiograph will be taken, using the customized x-ray tray.
  Interventions: Procedure: Early Implant Loading

INTERVENTIONS:
Procedure: Immediate Implant Loading — A single implant crown will be mounted on the implant immediately after implant placement
  Arms: Immediate Implant Loading
Procedure: Early Implant Loading — A single implant crown will be mounted on the implant 4 weeks after implant placement.
  Arms: Early Implant Loading

SUMMARY:
The planned study is designed to provide evidence for the application of early implant placement with partial bone-healing and either an immediate or an early restoration/ loading protocol.

Materials and methods

The study will be conducted according to the recommendations published as the CONSORT statement and respecting the intention to treat principle. Participants will be enrolled if they present with a mandibular first molar that has to be extracted, and require implant treatment for replacement of the molar. Ridge preservation using a well-documented xenogeneic bone substitute will be done following the extraction. After 12 weeks of healing, a cone-beam computed tomography (CBCT) and a digital intraoral scan will be taken, followed by digital planning of the implant position and the additive construction of a surgical drill guide by means of rapid prototyping using a 3-D printer. Afterwards, the participants will be randomized into the two study groups:

Group A (immediate loading): A screw-retained PMMA implant provisional bonded to a titanium base will be fabricated subtractively by computer aided design/ computer aided manufacturing (CAD/CAM), based on the data of the digitally planned implant position.

Group B (early loading): No further preparation has to be done.

Before finishing 16 weeks post-extraction, implants (Straumann Standard Implant RN, TiZr, minimum length: 10mm, minimum diameter 4.1mm) will be placed in both study groups using sCAIS. During surgery, the surgeon will not know if the participant was allocated to Group A or Group B. Directly after surgery, digital intraoral scans will be obtained, to record the final implant position. Afterwards, either the prepared implant provisional (Group A; immediate loading) or a healing cap (Group B, early loading) will be inserted into the implant.

4 weeks after implant placement the participants in Group B will receive a loaded, screw-retained implant provisional, based on the data of the post-surgery scan. 6-months after implant placement participants will receive final screw-retained single implant crowns. The study end will be a final follow-up visit after 12 months. Participants will be invited for further follow-up visits up to 5 years. (not part of the present proposal) Implant survival/ success will be evaluated according to the criteria described by Buser et al. All secondary outcomes will be assessed by validated indices and instruments.

DETAILED DESCRIPTION:
The planned study is designed to provide evidence for the application of early implant placement with partial bone-healing and either an immediate or an early restoration/ loading protocol.

Materials and methods

The study will be conducted according to the recommendations published as the CONSORT statement and respecting the intention to treat principle. Participants will be enrolled if they present with a mandibular first molar that has to be extracted, and require implant treatment for replacement of the molar. Ridge preservation using a well-documented xenogeneic bone substitute will be done following the extraction. After 12 weeks of healing, a cone-beam computed tomography (CBCT) and a digital intraoral scan will be taken, followed by digital planning of the implant position and the additive construction of a surgical drill guide by means of rapid prototyping using a 3-D printer. Afterwards, the participants will be randomized into the two study groups:

Group A (immediate loading): A screw-retained PMMA implant provisional bonded to a titanium base will be fabricated subtractively by computer aided design/ computer aided manufacturing (CAD/CAM), based on the data of the digitally planned implant position.

Group B (early loading): No further preparation has to be done.

Before finishing 16 weeks post-extraction, implants (Straumann Standard Implant RN, TiZr, minimum length: 10mm, minimum diameter 4.1mm) will be placed in both study groups using sCAIS. During surgery, the surgeon will not know if the participant was allocated to Group A or Group B. Directly after surgery, digital intraoral scans will be obtained, to record the final implant position. Afterwards, either the prepared implant provisional (Group A; immediate loading) or a healing cap (Group B, early loading) will be inserted into the implant.

4 weeks after implant placement the participants in Group B will receive a loaded, screw-retained implant provisional, based on the data of the post-surgery scan. 6-months after implant placement participants will receive final screw-retained single implant crowns. The study end will be a final follow-up visit after 12 months. Participants will be invited for further follow-up visits up to 5 years. (not part of the present proposal) Implant survival/ success will be evaluated according to the criteria described by Buser et al. All seconda

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Willingness to sign informed consent and to participate in the study
* Plaque index according to Silness and Loe of < 35% [26]

At site level:

* Presence of a mandibular first molar that has to be extracted
* Sufficient vertical interocclusal space for the placement of an implant crown (7 mm)
* Presence of an opposing natural or artificial tooth
* Ridge height sufficient for the placement of a ≥ 10 mm-long implant
* Sufficient ridge width for the placement of a 4.1mm diameter implant

Exclusion Criteria:

At patient level:

* Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance to the protocol
* Any disorder that would interfere with wound healing or represent a contraindication for implant surgery such as, but not limited to, uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates
* Pregnancy or lactation
* Heavy smoking habit with ≥ 10 cig/d
* Severe bruxism or clenching habits, present oro-facial pain at site level
* Insufficient ridge width/height for the study implant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival/success | 1 year
  An implant that is still in place 1 year after placement will be considered surviving. Implant success and survival rate will be defined according to established criteria : A surviving implant is defined as an implant in place at the time of the follow-up. A particular implant will be deemed a success if all of the following success criteria apply: Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (e. g. painful sensation) . Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics) . Absence of implant mobility on manual palpation . Absence of any continuous peri-implant radiolucency

SECONDARY OUTCOMES:
Prosthetic Success/ survival | 1 year
  During the prosthodontic examination, the implant supported prostheses will be examined for any complications and failures. Possible complications are: loss of retention , fracture and/or chipping, loosening of occlusal screw , fracture of occlusal screw , loosening of abutment , fracture of abutment. Prosthetic success is defined as the non-occurrence of any complications. If any complication occurs, but the crown is still in place, it will be considered surviving.
Accuracy of guided surgery | 1 year
  The accuracy of the final- compared to the digitally planned implant position, will be measured according to a previously conducted study at the University of Bern. Standard tessellation language (STL) files of the post-surgical implant scan will be imported into the coDiagnostiX software containing the previous digital plan. Treatment evaluation feature will be used to compare pre-planned to post-surgical implant positions. Virtually planned and postoperative implant STL files will be superimposed using the same occlusal/incisal surfaces of teeth as a reference. Angular and 3D deviation at implant crest and implant apex will be measured. The measurements will be performed by two independent examiners unaware of the treatment modalities.
Patient satisfaction | 1 year
  Patient satisfaction will be evaluated by means of a 10mm visual analogue scale (VAS) based questionnaire, which is administered after training the participant in using this form of scale. The evaluated items of the questionnaire will be the ease of cleaning, general satisfaction, comfort, aesthetics, stability, chewing ability and function.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abou-Ayash, PD Dr., Principal Investigator — University of Bern
Locations (1):
- Department of Reconstructive Dentistry, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data may be made available upon request.